CLINICAL TRIAL: NCT02990260
Title: Effect of Saccharomyces Cerevisiae in LDL Cholesterol
Acronym: HONEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lesaffre International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2016-A011094-47
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Live Saccharomyces cerevisiae (Active Comparator): Live Saccharomyces cerevisiae. 2 capsules per day (1 g).
  Interventions: Dietary Supplement: Saccharomyces cerevisiae
- Yeast cell wall (Active Comparator): Yeast cell wall. 2 capsules a day (700 mg).
  Interventions: Dietary Supplement: Lynside Wall Basic
- Placebo (Placebo Comparator): Maize starch and magnesium stearate. 2 capsules a day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Saccharomyces cerevisiae — Live Saccharomyces cerevisiae
  Arms: Live Saccharomyces cerevisiae
Dietary Supplement: Lynside Wall Basic — yeast cell walls
  Arms: Yeast cell wall
Dietary Supplement: Placebo — Maize starch and magnesium stearate
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effect of the consumption of a food supplement (live saccharomyces cerevisiae) on lipidic profile in moderate hypercholesterolemic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Moderate hypercholesterolemia (LDL cholesterol between 1.3 and 1.9 g/L) with maximum 1 associated cardiovascular risk factor.

Exclusion Criteria:

* Total cholesterol > 3.5 g/L (on an empty stomach)
* Triglycerides > 3 g/L (on an empty stomach)
* Familial hypercholesterolemia (IIa type)
* Diabete mellitus treated or not
* Subjects having consumed drugs known for their impact on lipid metabolism (statines, ezetimibes, colestyramin, fibrate...) in the month before beginning if the study and/or susceptible to consume such drugs during the study
* Subjects having consumed food supplements or functional foods known for their impact on cholesterolemia (phytosterols, phytostanols, policosanols, beta-glucans...) in the month before the study and/or susceptible to consume such products during the study
* Subjects having consumed probiotics food supplements in the month before the study and/or susceptible to consume such products during the study
* Subjects following a low diet regimen (intakes < 1500 kcal/day) in the month before the study and/or susceptible to start such a regimen during the study
* Food behaviour disorders diagnosed
* Subjects with rare serious diseases (rare digestive diseases, renal failure, cardiovascular diseases, tumor...) or having endure a serious surgery
* Subjects having endure bariatric surgery or having a gastric bypass in place
* Pregnant or lactating women
* Women willing a pregnancy Excessive alcohol consumption
* Susceptible to modify their tobacco consumption before the end of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-12; Primary Completion 2017-11 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Plasma LDL cholesterol | 8 weeks

SECONDARY OUTCOMES:
LDL cholesterol | 4 weeks
Total cholesterol | 4 weeks, 8 weeks
Triglycerides | 4 weeks, 8 weeks
HDL cholesterol | 4 weeks, 8 weeks
Apo B | 4 weeks, 8 weeks
Apo A1 | 4 weeks, 8 weeks
gamma GT | 4 weeks, 8 weeks
ASAT | 4 weeks, 8 weeks
ALAT | 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Pasteur de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided